CLINICAL TRIAL: NCT04452799
Title: Randomized Double-blind Controlled Parallel Study of (Hesperidin and Diosmin Mixture) for Treatment of COVID-19 Newly Diagnosed Patients in Egypt
Brief Title: Hesperidin and Diosmin for Treatment of COVID-19
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Prof. Dr. Kamal Mohammed Okasha, Professor, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1111
Record Dates: First submitted 2020-06-29; First posted 2020-06-30 (Actual); Last update posted 2020-06-30 (Actual); Status verified 2020-06

CONDITIONS: Coronavirus Infection
MeSH Terms: conditions — Coronavirus Infections | interventions — Hesperidin

STUDY DESIGN:
Intervention Model Description: Randomized double-blind controlled Parallel study
Who Masked: Participant, Care Provider
Masking Description: Randomized double-blind controlled Parallel study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- expermintal (Experimental): 1000mg of (Hesperidin and Diosmin mixture) three times daily for 7 days 1000mg of (Hesperidin and Diosmin mixture) two times daily for 3 days
  Interventions: Drug: Hesperidin and Diosmin mixture
- standard (Active Comparator): standard care therapy in quarantine hospitals
  Interventions: Drug: Hesperidin and Diosmin mixture

INTERVENTIONS:
Drug: Hesperidin and Diosmin mixture — Interventional Clinical Trial

SUMMARY:
SARS-CoV-2 or COVID-19 is representing the major global burden that implicated more than 10 million infected cases and 500 thousand deaths worldwide. The prevalence of this pandemic disease is expected to rise every day. The challenge is to control its rapid spread meanwhile looking for a specific treatment to improve patient outcomes. Hesperidin is a classical herbal medicine used worldwide for a long time with an excellent safety profile. Hesperidin is a well-known herbal medication used as an antioxidant and anti-inflammatory agent. Available shreds of evidence support the promising use of hesperidin in prophylaxis and treatment of COVID 19. Herein, we discuss the possible prophylactic and treatment mechanisms of hesperidin based on previous and recent findings. Hesperidin can block coronavirus from entering host cells through ACE2 receptors which can prevent the infection. Anti-viral activity of hesperidin might constitute a treatment option for COVID-19 through improving host cellular immunity against infection and its good anti-inflammatory activity may help in controlling cytokine storm. Hesperidin mixture with diosmin co-administrated with heparin protect against venous thromboembolism which may prevent disease progression. Based on that, hesperidin might be used as a meaningful prophylactic agent and a promising adjuvant treatment option against SARS-CoV-2 infection.

DETAILED DESCRIPTION:
Research Background and Rationale At the end of December 2019, pneumonia of unknown origin was detected in the hospitals of Wuhan city, China, and reported to the WHO country office for the first time [1-3]. After a few days, the Chinese government has confirmed the human-to-human transmission of the new infectious respiratory disease [4]. At the end of January 2020, the WHO declared the outbreak of severe acute respiratory syndrome (SARS), caused by a novel coronavirus (SARS-CoV-2), as an international public health emergency. The disease termed coronavirus 19 (COVID-19) rapidly transmitted from China to all over the world and subsequently the WHO declared it a global pandemic disease. The virulent virus structure is closely related to (SARS-CoV) strain with a single-stranded positive-sense RNA composition[5].

This pandemic disease is particularly of major importance to the whole world and especially to countries with a heavy population like Egypt. There is a critical need for emergent, continuous, and cost-effective health care delivery to infected people. Early detection and strategies for prevention of progression of COVID-19 would make a major difference for infected patients and would also be economically beneficial for a resource-constrained country.

People infected with COVID-19 may have no symptoms but still, act as a source of infection to other surrounding persons. The most common clinical manifestations following infection range from mild symptoms of (generalized fatigue, dry cough, low-grade fever, and sore throat) to severe symptoms of (typical severe acute respiratory distress syndrome (ARDS) and pneumonia)[6]. Although the tremendous scientific research effort is focusing mainly on the use of antiviral drugs, certain drug repurposing, and vaccine production for the treatment of COVID-19 patients, there is no specific cure or vaccine for treatment up till now. New drug development is a time-consuming process so that drug repositioning may be the optimum solution to control this pandemic infection.

Selected Drugs Hesperidin is a common flavone glycoside found in citrus fruit such as lemons and sweet oranges[7, 8]. Hesperidin has several pharmacological activities such as anti-atherogenic, antihyperlipidemic, antidiabetic, venotonic, cardioprotective, anti-inflammatory, and antihypertensive actions. The anti-inflammatory activity of hesperidin was mainly attributed to its antioxidant defense mechanism and suppression of pro-inflammatory cytokine production[7]. Hesperidin exhibited anti-viral activity against the influenza virus through a significant reduction of virus replication. Treatment of infected cells with hesperidin enhanced cell-autonomous immunity via activation and upregulation of p38 and JNK expression which is essential for cell defense mechanisms against influenza virus[9].

Hesperidin has been used as an herbal medicine for a long time. The safety of hesperidin was confirmed by FASEB (Federation of American Societies of Experimental Biology) upon request of the FDA. Toxicity studies have confirmed the high safety profile of hesperidin after oral intake. Results from oral toxicity studies showed the absence of adverse side effects after oral hesperidin ingestion of more than 2g /kg [10].

Daflon 500 mg is a marketed tablet dosage form containing a micronized flavonoid mixture of 50 mg of hesperidin and 450 mg of diosmin which used as vasoprotective venotonic agent[10]. This hesperidin mixture is characterized by its high safety profile. Continues oral administration for hesperidin mixture to rats for 13 and 26 weeks, using a very high dose of 35-fold of the daily dosage showed no toxicity with a high LD50 value of more than 3 g/kg body weight. Clinical trials used more than 2850 patients treated with the hesperidin mixture for a period of 6 weeks to 1 year showed normal hematological parameters, hepatic and renal functions with no signs of toxicity[11].

Hesperidin role in prevention and treatment of COVID 19 was recently published by our research team in Medical Hypotheses journal [12].

Unraveling host cellular receptors used for cellular entry of COVID-19 will provide possible lines for attack. Cell entry of COVID-19 depends on two consecutive steps, firstly binding of the viral spike (S-protein) to host cellular receptors followed by priming of S-protein by cell proteases. Recently, researchers showed that COVID-19 uses the ACE-2 receptor for entry [13] and the serine protease TMPRSS2 for priming of S-protein. Camostat mesylate, a serine protease inhibitor drug blocked virus entry and was used as a COVID-19 treatment in Japan[14].

COVID-19 binds to the ACE-2 receptor through its specific Spike-receptor binding domain (RBD) sequence to form the SARS-CoV-2-RBD-ACE-2 complex. The proposed computational activity of 78 anti-viral drugs against the human ACE2 receptor was screened using homology modeling. This study showed that hesperidin is the only compound that could target the binding interface between SARS-CoV-2 Spike and ACE2 human receptors. based on virtual screening, hesperidin may disrupt the interaction of ACE2 with RBD of SARS-CoV-2 thus block its entry into the lung cells [15]. Therefore, hesperidin can be used as a promising prophylactic agent against COVID-19 infection.

Host antiviral responses against COVID-19 infection depend on the activation of both the immune systems and cellular self-defense mechanisms. Immunity plays a major role in the protection of the host against viral infection. The occurrence of immune over-response or immune deficiency is responsible for the condition of infected patients becoming critical or severe[16]. The anti-viral activity of hesperidin against the influenza virus involves its role in the activation of the mitogen-activated protein kinase (MAPK) pathway. The MAPK host defense cascade contributes to efficiently restraining viral replication, spread, and minimizing tissue damage[9]. A recent study showed that the interferon-MAPK pathway played an important role in the COVID-19 immune response[16]. Therefore, hesperidin by its activation to host immunity my help against COVID-19 viral replication and hence its progression which will improve the patient outcome.

Patients infected with COVID-19 exhibited what is called "cytokine storm" which initiated primarily as an inflammatory response and resulted in uncontrolled over-production of soluble markers of inflammation. Available evidence showing that cytokine storm, is a major cause for the development of ARDS. Cytokine storm involves the release of various immune-active molecules such as Interferons (e.g. IFNγ), interleukins (e.g. IL-1β, IL-2, IL-6), chemokines, and tumor necrosis factor-alpha (TNF-α ) [17].

Hesperidin with its high anti-inflammatory activity inhibited the secretion of pro-inflammatory cytokines such as IFN-γ and IL-2[18]. Besides, hesperidin inhibited IL 1β stimulated inflammatory responses by inhibiting the activation of the NF κB signaling cascade[19]. It also played a major rule in suppressing the release of inflammatory markers such as (TNFα and IL-6) in type 2 diabetic patients[20]. Therefore, it can be used as adjuvant therapy to control the severe inflammatory reaction against COVID-19.

Activation of coagulation pathways following the immune response to COVID-19 infection promotes clot formation. The proposed mechanism of formation of micro thrombosis involves the occurrence of procoagulant-anticoagulant imbalance, platelet activation, and converting fibrinogen to fibrin. Disseminated intravascular coagulation predisposes to the development of multiorgan failure especially in severe infected cases[21].

A prophylactic dose of heparin (with low molecular weight, LMWH) is recommended for protection against venous thromboembolism in COVID-19 hospitalized patients[21]. In this context, it is essential to highlight the role of concomitant administration of hesperidin and diosmin mixture with heparin for protection against thromboembolism. Results from previous clinical trials that used Daflon 500 mg with LMWH confirmed the significant effect of this combination compared to LMWH alone in preventing the incidence of pulmonary embolism and deep vein thrombosis. Therefore, co-administration of LMWH and Daflon 500 mg can significantly inhibit clot formation and prevent disease progression [22].

Diagnostic criteria The viral research institution in China has conducted preliminary identification of the SARS-CoV-2 through the classical Koch's postulates and observing its morphology through electron microscopy[1]. So far, the golden clinical diagnosis method of COVID-19 is nucleic acid detection in the nasal and throat swab sampling or other respiratory tract samplings by real-time PCR and further confirmed by next-generation sequencing Clinical classification of patients Patients can be grouped into three categories: asymptomatic, upper respiratory tract infection (URTI) when presenting with rhinitis, pharyngitis, or isolated low-grade fever and myalgia, and lower respiratory tract infections (LRTI) when presenting with symptoms of pneumonia or bronchitis[3].

Side effects of (Hesperidin and Diosmin mixture, Daflon®) Like all medicines, Daflon 500 mg can cause side effects, although not everybody gets them. Some cases of commonplace gastrointestinal disorders and neurovegetative disorders (feeling of discomfort) have been described, which do not require stopping the treatment.

Safety concerns of (Hesperidin and Diosmin mixture, Daflon®) Daflon 500 mg tablets is POSSIBLY SAFE for most people when taken by mouth for up to 6 months. The safety of using it for a longer period of time is unknown. Side effects include stomach pain and upset, diarrhea, and headache.

Contraindications of (Hesperidin and Diosmin mixture, Daflon®) No reported contraindications.

Interactions of (Hesperidin and Diosmin mixture, Daflon®) No sever drug-drug interactions, only moderate and minor interactions

* Celiprolol: (Moderate drug-drug interaction) Hesperidin may reduce the absorption of celiprolol.
* Diltiazem: (Moderate drug-drug interaction) Hesperidin may reduce the absorption of diltiazem.
* Verapamil: (Moderate drug-drug interaction) Hesperidin may increase the absorption of verapamil.
* Antihypertensive drugs: (Moderate drug-drug interaction) Hesperidin may lower high blood pressure might cause your blood pressure to go too low.
* Anticoagulant / Antiplatelet drugs: (Moderate drug-drug interaction) Hesperidin may slow blood clotting which might increase the chances of bruising and bleeding.
* Sedative medications (Benzodiazepines) (Moderate drug-drug interaction) Hesperidin may cause too much sleepiness.

Special Precautions & Warnings:

* Pregnancy and breast-feeding: Hesperidin is POSSIBLY SAFE for pregnant or breast-feeding women when taken by mouth with diosmin.
* Bleeding disorder: Hesperidin might slow blood clotting and increase the risk of bleeding. In theory, hesperidin might make bleeding disorders worse.
* Low blood pressure: Hesperidin might lower blood pressure. In theory, taking hesperidin might make blood pressure become too low in people who already have low blood pressure.
* Surgery: Hesperidin might prolong bleeding. There is concern that hesperidin might increase the risk of bleeding during and after surgical procedures. Stop taking hesperidin at least 2 weeks before a scheduled surgery.

Research Objectives

This research proposal was employed as a practical strategy for providing a suitable drug or drug combination for possible treatment of COVID-19 infected patients. This drug may help to prevent the progression of respiratory complications. This can be achieved through different goals as following:

1. Screening of different drugs related to different pharmacological classes depending on its possible activity against COVID-19 virus.
2. Providing cost-effective and easy-to-implement treatment strategy for infected patients and/or patients with high risk of developing respiratory failure.
3. Finally, this clinical strategy remains an important goal in improving Egyptian health state which can save their life meanwhile save a lot of money.

Scope of Work The scope of work will be conducted through

1. Use of newly repurposed drug (Daflon 500 mg) for treatment of COVID-19 infected people.
2. Evaluation of the effect of the drug on the symptomatic treatment of mild COVID-19 patients through a clinical trial designed according to WHO (Clinical management of severe acute respiratory infection (SARI) when COVID-19 disease is suspected) interim guidance published at 13 March 2020.
3. Investigating the impact of the drug on the prevention of sever compilations such as Acute Respiratory Distress Syndrome (ARDS).

Randomized double-blind controlled Parallel study of (Hesperidin and Diosmin mixture, Daflon®) for treatment of Covid-19 newly diagnosed Patients in Egypt.

Study design This study will be a double blind randomized controlled parallel study Study population and Methods Setting This study will be on Patients currently being granted at designated hospitals affiliated to Ministry of Higher Education. Patients will be randomized to either receive Daflon versus control group who will receive standard care Patients Hospitalized patients with confirmed COVID-19 will included in this study according to the following criteria; Adult (18-65 Years old), both sexes, PCR positive in nasopharyngeal sample at admission. In addition, inclusion criteria will involve newly diagnosed asymptomatic or with upper respiratory tract infection (URTI) patients who will present with rhinitis, pharyngitis, or isolated low-grade fever and myalgia.

Informed consent Before being included in the study, patients meeting inclusion criteria will give their written informed consent to participate to the study. An information document that clearly indicates the nature of the study and the risks or side effects and the benefits associated with the participation to the study will be given to each participant. The study will be conducted in accordance with the Ethical standards of Helsinki Declaration. The protocol will be submitted to the National Ethic Committee for reviewing and approval. This trial will be registered as Clinical Trial.

Procedure Patients will be seen at baseline for enrolment, initial data collection and treatment at day-0. The follow up duration will be 28 days or till PCR negative. Starting from day 1, each day, patients will receive standardized care or Daflon 1000 mg, three times daily for 10 days. Symptomatic treatment and antibiotics as a measure to prevent bacterial superinfection will be provided based on clinical judgment for all participants. All participants will be submitted to blood samples collection at base line and after the follow up period for RT- PCR assay and to evaluate the change in serum IL1β, TNF-α, hsCRP. CBC will be done for Lymphocyte count. Changes in respiratory rate and PaO2 will be assessed. Furthermore, mortality rate will be calculated.

Outcomes Primary Outcome Measures: is RT-PCR negative Secondary Outcome Measures include: changes in respiratory rate and PaO2, change in serum IL1β, TNF-α, hsCRP, Lymphocyte count, mortality rate and occurrence of side-effects.

Randomized double-blind controlled Parallel study of (Hesperidin and Diosmin mixture, Daflon®) for treatment of Covid-19 newly diagnosed Patients in Egypt.

Study design: Randomized double-blind controlled Parallel study Study Type: Interventional Clinical Trial Enrolment: 50 participants in each arm Allocation: Randomized Assignment: Parallel Intervention Model Description: Two parallel groups randomly asserted Masking: Double (Participant, Investigator) Primary Purpose: Treatment or efficacy plus safety Estimated Study Start Date: 01/07/2020 Estimated Primary Completion Date: 15/07/2020 Estimated Study Completion Date: 01/10/2020 Arms

Experimental:

1000mg of Daflon three times daily for 10 days

Active Comparator:

Standard care delivered in the isolation hospitals. Outcomes

Primary Outcome Measures:

PCR negative

Secondary Outcome Measures:

Changes in respiratory rate Change in patients PaO2 Change in serum IL1β Change in serum TNF-α Change in serum hsCRP CBC for Lymphocyte count Reported side effects Mortality rate

Inclusion Criteria:

Confirmed cases of Covid-19 (all by RT-PCR) Newly diagnosed asymptomatic or with upper respiratory tract infection (URTI) patients who will present with rhinitis, pharyngitis, or isolated low-grade fever and myalgia, Adult (18-65 Years old) Both sexes

Exclusion Criteria:

Patients with bleeding disorders Patients with low to very low blood pressure Patients after surgery Immunocompromised patients taking medication upon screening

ELIGIBILITY:
Inclusion Criteria:

Confirmed cases of Covid-19 (all by RT-PCR) Newly diagnosed asymptomatic or with upper respiratory tract infection (URTI) patients who will present with rhinitis, pharyngitis, or isolated low-grade fever and myalgia, Adult (18-65 Years old) Both sexes

Exclusion Criteria:

Patients with bleeding disorders Patients with low to very low blood pressure Patients after surgery Immunocompromised patients taking medication upon screening

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-07-01 (Estimated); Primary Completion 2020-10-01 (Estimated); Study Completion 2020-10-30 (Estimated)

PRIMARY OUTCOMES:
PCR test | 14 days
  PCR negative

SECONDARY OUTCOMES:
respiratory rate | 14 days
  Changes in respiratory rate
patients PaO2 | 14 days
  Change in patients PaO2
serum IL1β | 14 days
  change in serum IL1β
serum TNF-α | 14 days
  changes in serum TNF-α
Mortality rate | 14 days
  decrease in Mortality rate

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Haggag YA, El-Ashmawy NE, Okasha KM. Is hesperidin essential for prophylaxis and treatment of COVID-19 Infection? Med Hypotheses. 2020 Nov;144:109957. doi: 10.1016/j.mehy.2020.109957. Epub 2020 Jun 6. PMID 32531538